CLINICAL TRIAL: NCT06555458
Title: The Effect of Sedation on Rebound Pain in Knee Arthrplasty Performed Under Spinal Anesthesia
Brief Title: The Effect of Sedation on Rebound Pain in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E1-23-4142
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Total Knee Arthroplasty; Sedation
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients will receive the standardized pre-op meds and spinal anesthetic.
  Once the patient's spinal is performed, patient will receive the following:
  Start with bolus of 0.4 microgram/kg over 10 minutes, and then infusion of 0.4 microgram/kg/hr infusion will be stopped after the last staple or suture is performed on the incision.
  Interventions:
  Drug: Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Saline (Placebo Comparator): Patients will receive the standardized pre-op meds and spinal anesthetic. Once the spinal anesthetic is performed,patient will receive the same infusion rates as in the Dexmedetomidine arm, however with Normal Saline as a Placebo.
  Interventions:
  Drug: Normal Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patient group to be given dexmedetomidine
  Arms: Dexmedetomidine
Drug: Saline — Patient group to be given salin
  Arms: Saline

SUMMARY:
Dexmedetomidine is often used for sedation procedures. It has also been shown to have a pain-protective effect. Researchers predicted that using dexmedetomidine for sedation in total knee arthroplasties performed under spinal anesthesia would reduce the frequency of rebound pain and pain scores.

DETAILED DESCRIPTION:
Randomization will take place before the patient enters the operating room. After spinal anesthesia is applied, 0.4 mcg/kg sedadomide loading will be done for 10 minutes in the sedation group, and then 0.4 mcg/kg/h sedadomide infusion will continue until the end of the surgery. Patients selected for the control group will be given the same amounts of saline. At the end of the surgical procedure, saline and sedadomide infusions will be stopped. All patients will undergo an adductor canal block under USG guidance in the recovery room. 50 mg of buvacin will be given to the block area. Patients will be fitted with a patient control analgesia device, which only provides bolus application and provides 20 mg of madol in each bolus. Postoperatively, sudden onset severe withdrawal pain outside the normal course of pain starting within 48 hours will be followed and Vas-bromage monitoring will be done at 0, 1, 2, 4, 8, 12, 24, 36, 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee arthroplasty American Society of Anesthesiologist score of 1-3 Age 18-85 Elective total knee arthroplasty under spinal anesthetic.

Exclusion Criteria:

* Situations in which spinal anesthesia is contraindicated
* Advanced organ failure states(cardiac,hepatic,respiratuar or renal)
* Pregnancy
* BMI > 40 kg/m^2
* Do not want to participate in the study
* Younger than 18 or older than 85
* Have bilateral total knee arthroplasty or resurgery
* Develop an unexpected intraoperative surgical complication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Rebound pain VAS scores and incidence of rebound pain | 48 hours after surgery
  Rebound pain-defined as transient acute postoperative pain within 12-24hrs that ensues following resolution of sensory blocked.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, ÇANKAYA, Turkey (Türkiye)